CLINICAL TRIAL: NCT04351269
Title: Retrospective Experience of CIED Implantation With Piedmont Athens Regional Electrophysiology
Brief Title: Retrospective Experience Of CIED Implantation
Status: Completed | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CPR-2212
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Results first posted 2022-05-18 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Cardiac Disease; Heart Failure; Coronary Artery Disease
MeSH Terms: conditions — Heart Diseases; Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- CanGaroo Envelope: Patients who received a CanGaroo Envelope with their Cardiac Implantable Electronic Device (CIED) implantation.
  Interventions: Device: CanGaroo Envelope
- TYRX Envelope: Patients who received a TYRX Envelope with their Cardiac Implantable Electronic Device (CIED) implantation.
  Interventions: Device: TYRX Envelope
- No Envelope: Patients who had their Cardiac Implantable Electronic Device (CIED) implanted with no envelope.

INTERVENTIONS:
Device: CanGaroo Envelope — CanGaroo Envelope with Cardiac Implantable Electronic Device (CIED) implantation
  Groups: CanGaroo Envelope
Device: TYRX Envelope — TYRX Envelope with Cardiac Implantable Electronic Device (CIED) implantation
  Groups: TYRX Envelope

SUMMARY:
The objective of this study is to retrospectively gather information on patients who underwent a CIED procedure with either a CanGaroo Envelope, TYRX Envelope, or no envelope.

DETAILED DESCRIPTION:
A single center will retrospectively review up to 700 subjects who underwent implantation of a CIED with a CanGaroo Envelope, TYRX Envelope, or no envelope. All sets of subjects enrolled will also be examined for any follow-up visits and/or adverse events that occurred up to 12 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any patient that had a CIED implanted with either a CanGaroo Envelope, a TYRX Envelope, or no envelope on or after March 27, 2017

Exclusion Criteria:

* Any patient that had a CIED implanted with any other type of envelope
* Any patient that had a CIED implanted prior to March 27, 2017

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients who underwent a CIED implantation utilizing a CanGaroo Envelope hydrated in saline, a CanGaroo Envelope hydrated in an antibiotic solution, a TYRX Envelope, or no envelope.
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Riebman, MD, Study Director — Aziyo Biologicgs, Inc.
Locations (1):
- Piedmont Athens Electrophysiology, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CanGaroo Envelope | TYRX Envelope | No Envelope
Started | 237 | 260 | 100
Completed | 165 | 219 | 71
Not Completed | 72 | 41 | 29
Not completed — Subjects did not meet Inclusion criteria after protocol revision B | 70 | 32 | 29
Not completed — CanGaroo Envelope used during a previous procedure | 0 | 1 | 0
Not completed — Subjects had both CanGaroo Envelope and TYRX Envelope used during procedure | 1 | 1 | 0
Not completed — Subjects followed long-term at different health care system | 0 | 4 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- CanGaroo Envelope: Patients who received a CanGaroo Envelope with their CIED implantation.
  CanGaroo Envelope: CanGaroo Envelope with CIED implantation
- TYRX Envelope: Patients who received a TYRX Envelope with their CIED implantation.
  TYRX Envelope: TYRX Envelope with CIED implantation
- No Envelope: Patients who had their CIED implanted with no envelope.
- Total: Total of all reporting groups
Arm/Group | CanGaroo Envelope | TYRX Envelope | No Envelope | Total
Number analyzed (Participants) | 165 | 219 | 71 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (13.2) | 70.3 (13.5) | 74.2 (11.0) | 72.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 79 | 24 | 167
  Male | 101 | 140 | 47 | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 3
  Not Hispanic or Latino | 159 | 206 | 68 | 433
  Unknown or Not Reported | 6 | 10 | 3 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 16 | 20 | 3 | 39
  White | 143 | 183 | 64 | 390
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 5 | 12 | 4 | 21
BMI, Continuous [Mean (Standard Deviation); unit: kg/m²] | 28.6 (6.5) | 30.6 (7.2) | 31.0 (6.3) | 29.9 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Infection Post Procedure
Description: Major CIED infections are defined as a CIED infection resulting in one or more of the following:
  * CIED system removal
  * Any invasive procedure (e.g., pocket opened) without system removal
  * Treatment with antibiotic therapy if the subject is not a candidate for system removal and infection recurrence after completion of antibiotic therapy or evidence of deep infection with wound dehiscence, erosion, or purulent drainage
  * Death
Time Frame: 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | CanGaroo Envelope | TYRX Envelope | No Envelope
Number analyzed (Participants) | 165 | 219 | 71
Participants | 2 | 0 | 0

2. Secondary Outcome: Number of Participants With Pocket Related Issues Prompting an Office Visit
Description: Any pocket related issues that prompted an office visit
Time Frame: 12 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | CanGaroo Envelope | TYRX Envelope | No Envelope
Number analyzed (Participants) | 165 | 219 | 71
Participants
  Hematoma | 2 | 2 | 0
  Pocket Infection | 2 | 0 | 0
  Lead Dislodgement | 1 | 3 | 0
  Site Drainage | 1 | 0 | 0
  Thrombosis | 1 | 0 | 0
  Superficial Surgical Site Infection (SSI) | 1 | 2 | 0
  Lead Revision | 0 | 1 | 0
  Hemothorax | 0 | 1 | 0
  Erythema & Fever | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 12 months post-procedure
Arm/Group | CanGaroo Envelope | TYRX Envelope | No Envelope
All-Cause Mortality (participants affected / at risk) | 0/165 | 10/219 | 0/71
Serious Adverse Events (participants affected / at risk) | 9/165 | 7/219 | 1/71
Other Adverse Events (participants affected / at risk) | 0/165 | 0/219 | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CanGaroo Envelope (N=165) | TYRX Envelope (N=219) | No Envelope (N=71)
Hematoma (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Pocket Infection (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Lead Dislodgement (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Superficial Surgical Site Infection (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Lead Revision (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hemothorax (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lead Perforation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The limitations of this study are its retrospective, observational nature, non-randomized design, limited duration of follow up, and single-physician design. The lack of randomization may introduce bias in the selection of patients for implantation with CIED envelopes and in the choice between CanGaroo and TYRX Envelopes. Finally, the duration of follow up may not have captured late adverse events, limiting data on longer-term outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT04351269/Prot_SAP_000.pdf